CLINICAL TRIAL: NCT03337178
Title: Fitbit Pilot Study to Increase Physical Activity and Overall Health in Post-operative Lumbar Degenerative Spinal Stenosis Patients
Brief Title: Fitbit Pilot Study in Post-operative Lumbar Degenerative Spinal Stenosis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The London Spine Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ReDA359
Record Dates: First submitted 2017-07-11; First posted 2017-11-08 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Lumbar Degenerative Spinal Stenosis

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Standard of care
- Blinded Fitbit (Experimental): Blinded Fitbit, no step goal, and no activity feedback
  Interventions: Behavioral: Blinded Fitbit
- Fitbit (Experimental): Fitbit plus step goal and activity feedback
  Interventions: Behavioral: Fitbit

INTERVENTIONS:
Behavioral: Blinded Fitbit — Fitbit is worn for 3 months post-operatively with no activity feedback or step goals
  Arms: Blinded Fitbit
Behavioral: Fitbit — Fitbit is worn for 3 months post-operatively with feedback and step goals
  Arms: Fitbit

SUMMARY:
Spinal stenosis is a common orthopedic spine condition that limits individuals ability to walk and stand because of nerve compression. Surgical treatment can alleviate leg pain and improve function such as increasing physical activity. This study will use Fitbit technology to monitor patient's post-operative physical activity. It will evaluate the efficacy of a Fitbit incentive based walking program on improving post-operative physical activity and rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age and older
* diagnosed with neurogenic claudication or radiculopathy secondary to central or lateral recess stenosis between L3-L5 confirmed by CT or MRI
* consent for surgical treatment

Exclusion Criteria:

* traumatic stenosis from a pathologic fracture
* inflammatory spine disease
* peripheral arterial disease
* hip or knee arthritis or pulmonary or circulatory diseases for which exercise is contraindicated
* severe or progressive neurologic deficit effecting ambulatory ability
* cancer
* no access to a computer or mobile device
* inability to complete the questionnaires or provide follow-up (i.e. lack of permanent address, substance abuse, interfering psychiatric illness).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-Paced Walking Test | Change in 3 months post-op from baseline
  Variability of the self-paced walking test

SECONDARY OUTCOMES:
Patient Recruitment | Number consented by 17 months
  Participants will be included if they are 60 years of age and older, diagnosed with neurogenic claudication or radiculopathy secondary to central or lateral recess stenosis between L3-L5 confirmed by CT or MRI, and consent for surgical treatment. Include patients with Grade 1 spondylolithesis. Patients will be excluded if the stenosis was not degenerative (i.e. traumatic stenosis from a pathologic fracture), they had inflammatory spine disease, they had peripheral arterial disease, or pulmonary or circulatory diseases for which exercise is contraindicated, osteoarthritis in the lower extremities, severe or progressive neurologic deficit requiring urgent surgery, cancer, previous lumbar surgery, they have no access to a computer or mobile device, an inability to complete the questionnaires or provide follow-up (i.e. lack of permanent address, substance abuse, interfering psychiatric illness).
Self-paced walking test | Change in 3 months post-op from baseline
  Self-paced walk test (SPWT) is a validated measure of walking capacity in lumbar degenerative spinal stenosis. The individual walks comfortably at his/her own pace until he/she must rest due to symptoms of back or leg pain. The total time and distance walked is recorded, time/distance to onset of symptoms, and nature and location of symptoms (pain numbness/tingling, weakness or fatigue), average walking speed, and reason for termination (symptoms of LSS, fatigue, shortness of breath, pain, other comorbidities). Patients are not permitted to use an assistive device. The test is either self-terminated (complete stop of 3 seconds or more) due to symptoms or at 30 minutes whichever occurs first. Participants are asked to indicate when they first experience symptoms.
Steps walked/day | Change in 3 months post-op from baseline
  Comparison of Fitbit activity data of steps taken between groups
Leg Pain | Change in 3 months post-op from baseline
  Numeric Rating Score for Leg Pain. The (NRS) for leg pain numeric rating scale ranges from 0 to 10, with lower scores indicating less severe symptoms
Back Pain | Change in 3 months post-op from baseline
  Numeric Rating Score for Back Pain. The (NRS) for back pain numeric rating scale ranges from 0 to 10, with lower scores indicating less severe symptoms
General Health | Change in 3 months post-op from baseline
  General health assessed by SF12. The SF12 is a generic, multidimensional self-report health questionnaire and is validated when applied to the spine patient. Questions are categorized into scales for general health, physical functioning, social functioning, role limitation-physical, role limitation-emotional, mental health, energy/fatigue, pain, comparative health. These are summarized into the SF12-physical component summary score (PCS) and mental component summary score (MCS). Scores range from 0 to 100. Higher scores imply better functioning.
Functional Ability | Change in 3 months post-op from baseline
  Functional ability assessed by Oswestry Disability Index. Oswestry Disability Index (ODI) is a validated questionnaire in lumbar degenerative spinal stenosis patients that assesses back pain-related disability. A higher score denotes worsening disability.
Functional Ability | Change in 3 months post-op from baseline
  Functional ability assessed by Swiss Spinal Stenosis Questionnaire. Swiss spinal stenosis questionnaire (SSS) is a validated 12-item condition-specific instrument for lumbar degenerative spinal stenosis that is known to be internally consistent and reliable and responsive to clinical change. It is a self-reported measure of pain and physical function. Higher scores represent worse physical function. The score for physical function was calculated as the un-weighted mean of the five items of the scale. The resulting possible scores of 1-4 represent mild to severe limitation in physical function. The Symptom Severity Scale will be used by averaging the scores the seven items. Responses range from 1-7 indicating mild to severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada